CLINICAL TRIAL: NCT02214433
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of Debio 1450 in Healthy Subjects
Brief Title: A Multiple Dose Study of Debio 1450 [Intravenous (IV) and Oral] in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Debio 1450-103; 217595 (Other: CRO); NCT02214355 (obsolete NCT alias)
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Bacterial Infections
Keywords: Antibiotic; Antibiotic Resistant Bacterial Infection
MeSH Terms: conditions — Bacterial Infections | interventions — Capsules; afabicin; Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- Part A Period 1 Debio 1450 IV Solution (Experimental): Part A Debio 1450 IV solution infused over two hours on Day 1 after fasting
  Interventions: Drug: Debio 1450 IV Solution
- Part A Period 2 Debio 1450 Tablet (Experimental): Debio 1450 Tablet oral dosing once on Day 5, after fasting
  Interventions: Drug: Debio 1450 Tablet
- Part A Period 3 Debio 1450 Tablet (Experimental): Debio 1450 Tablet oral dosing once on Day 9, 30 minutes after a high calorie, high fat breakfast, after fasting
  Interventions: Drug: Debio 1450 Tablet
- Part A Period 4 Debio 1450 Tablet (Experimental): After preparation with Pantoprazole, Pantoprazole taken with Debio 1450 Tablet oral dosing once on Day 14, after fasting
  Interventions: Drug: Debio 1450 Tablet; Drug: Pantoprazole
- Part B Placebo All Cohorts (Placebo Comparator): Placebo IV solution on days 1-5 and then Placebo Tablet or Capsule on Days 6-10, according to the cohort dosing schedule
  Interventions: Drug: Placebo IV Solution; Drug: Placebo Tablet or Capsule
- Part B Debio 1450 Cohort 1 (Experimental): Debio 1450 IV solution, once daily on days 1-5, then Debio 1450 Tablet, once daily on days 6-10
  Interventions: Drug: Debio 1450 IV Solution; Drug: Debio 1450 Tablet
- Part B Debio 1450 Cohort 2a (Experimental): Debio 1450 IV solution, once daily on day 1
  Interventions: Drug: Debio 1450 IV Solution
- Part B Debio 1450 Cohort 3 (Experimental): Debio 1450 IV solution, twice daily on days 1-5, then Debio 1450 Capsule, twice daily on days 6-10
  Interventions: Drug: Debio 1450 IV Solution; Drug: Debio 1450 Capsule
- Part B Debio 1450 Cohort 4 (Experimental): Debio 1450 IV solution, twice daily on days 1-5, then Debio 1450 Capsule, twice daily on days 6-10
  Interventions: Drug: Debio 1450 IV Solution; Drug: Debio 1450 Capsule
- Part B Debio 1450 Cohort 2b (Experimental): Debio 1450 IV solution, once daily on days 1-5, then Debio 1450 Capsule, once daily on days 6-10
  Interventions: Drug: Debio 1450 IV Solution; Drug: Debio 1450 Capsule
- Part C Debio 1450 (Experimental): Debio 1450 (IV formulation in Period 1, capsule formulation in Periods 2, 4 and 5 (with Pantoprazole), and Debio 1450 oral solution in Period 3).
  Interventions: Drug: Debio 1450 IV Solution; Drug: Debio 1450 Capsule; Drug: Debio 1450 Oral Solution; Drug: Pantoprazole

INTERVENTIONS:
Drug: Placebo IV Solution — A sterile IV solution of 5% dextrose in water
  Arms: Part B Placebo All Cohorts
Drug: Debio 1450 IV Solution — A white to off-white powder (40 mg Debio 1450 per vial) to be reconstituted and formulated in a sterile IV solution of 5% dextrose in water
  Arms: Part A Period 1 Debio 1450 IV Solution; Part B Debio 1450 Cohort 1; Part B Debio 1450 Cohort 2a; Part B Debio 1450 Cohort 2b; Part B Debio 1450 Cohort 3; Part B Debio 1450 Cohort 4; Part C Debio 1450
Drug: Placebo Tablet or Capsule — Placebo tablet or capsule, matching Debio 1450 coated tablet or capsule
  Arms: Part B Placebo All Cohorts
Drug: Debio 1450 Tablet — Debio 1450 40 mg coated tablets
  Arms: Part A Period 2 Debio 1450 Tablet; Part A Period 3 Debio 1450 Tablet; Part A Period 4 Debio 1450 Tablet; Part B Debio 1450 Cohort 1
Drug: Debio 1450 Capsule — Debio 1450 40 mg capsules
  Arms: Part B Debio 1450 Cohort 2b; Part B Debio 1450 Cohort 3; Part B Debio 1450 Cohort 4; Part C Debio 1450
Drug: Debio 1450 Oral Solution — Lyophilized Debio 1450 (40 mg per vial) reconstituted in 5% dextrose in water
  Arms: Part C Debio 1450
Drug: Pantoprazole — Pantoprazole 40 mg orally
  Arms: Part A Period 4 Debio 1450 Tablet; Part C Debio 1450

SUMMARY:
Debio 1450-103 is a trial to study the pharmacokinetics (PK) of an experimental drug called Debio 1450 in healthy adult volunteers. Originally, Part A was registered separately (in NCT02214355). The registrations have been revised so all parts of this single trial (Parts A-C) are now included in this single registration (NCT02214433).

The primary purpose of each part is provided below:

* 10 volunteers participate in PART A to assess the PK of a single oral dose of Debio 1450 (tablet formulation) under varying gastric conditions
* 40 volunteers participate in PART B to assess the safety, tolerability and PK of multiple ascending doses of Debio 1450, administered sequentially IV and orally, once or twice daily.
* An additional 10 volunteers participate in PART C which is designed to assess the absolute bioavailability of various formulations of Debio 1450 under varying gastric conditions

The dose administered during Part A is based on the safety, tolerability and PK data from study Debio 1450-102 [NCT02162199], a single ascending dose (SAD) study, in which single oral doses up to 800 mg/day are being investigated. Doses are adjusted during Parts B and C based on the available safety and PK data from preceding cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and/or contraception
* Is willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related to food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Has a history or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding)
  3. the analysis of results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinically significant change from baseline in safety parameters | within 10 days post-dose
  Categories: vital signs, 12-lead electrocardiogram (ECG), clinical laboratory parameters, adverse events, pulmonary function, physical examination, concomitant medication
Maximum observed plasma concentration (Cmax) of Debio 1450 (prodrug) and Debio 1452 (active moiety) | within 60 hours post-dose, depending on the assessment schedule for the cohort
  Categories: Placebo Tablet or Capsule, Placebo IV Solution, Debio 1450 IV solution, Debio 1450 Tablet, Debio 1450 Capsule, Debio 1450 oral solution
Time of maximum observed plasma concentration (tmax) of Debio 1450 and Debio 1452 | within 60 hours post-dose, depending on the assessment schedule for the cohort
  Categories: Placebo Tablet or Capsule, Placebo IV Solution, Debio 1450 IV solution, Debio 1450 Tablet, Debio 1450 Capsule, Debio 1450 oral solution
Area under the plasma concentration-time curve (AUC) of Debio 1450 and Debio 1452 | within 60 hours post-dose, depending on the assessment schedule for the cohort
  Categories: Placebo Tablet or Capsule, Placebo IV Solution, Debio 1450 IV solution, Debio 1450 Tablet, Debio 1450 Capsule, Debio 1450 oral solution
Percentage of AUC(0-o) that is due to extrapolation beyond the last quantifiable concentration measurement (%AUCex) of Debio 1450 and Debio 1452 | within 60 hours post-dose, depending on the assessment schedule for the cohort
  Categories: Placebo Tablet or Capsule, Placebo IV Solution, Debio 1450 IV solution, Debio 1450 Tablet, Debio 1450 Capsule, Debio 1450 oral solution
Elimination half-life (t1/2) of Debio 1450 and Debio 1452 | within 60 hours post-dose, depending on the assessment schedule for the cohort
  Categories: Placebo Tablet or Capsule, Placebo IV Solution, Debio 1450 IV solution, Debio 1450 Tablet, Debio 1450 Capsule, Debio 1450 oral solution
Terminal elimination rate constant (Az) of Debio 1450 and Debio 1452 | within 60 hours post-dose, depending on the assessment schedule for the cohort
  Categories: Placebo Tablet or Capsule, Placebo IV Solution, Debio 1450 IV solution, Debio 1450 Tablet, Debio 1450 Capsule, Debio 1450 oral solution
Mean residence time (MRT) of Debio 1450 and Debio 1452 | within 60 hours post-dose, depending on the assessment schedule for the cohort
  Categories: Placebo Tablet or Capsule, Placebo IV Solution, Debio 1450 IV solution, Debio 1450 Tablet, Debio 1450 Capsule, Debio 1450 oral solution
Apparent clearance following oral administration (CL/F) of Debio 1450 and Debio 1452 | within 60 hours post-dose, depending on the assessment schedule for the cohort
  Categories: Placebo Tablet or Capsule, Placebo IV Solution, Debio 1450 IV solution, Debio 1450 Tablet, Debio 1450 Capsule, Debio 1450 oral solution
Apparent volume of distribution of Debio 1450 and Debio 1452 during terminal phase (Vz/F) | within 60 hours post-dose, depending on the assessment schedule for the cohort
  Categories: Placebo Tablet or Capsule, Placebo IV Solution, Debio 1450 IV solution, Debio 1450 Tablet, Debio 1450 Capsule, Debio 1450 oral solution
Cumulative amount of unchanged Debio 1450 and Debio 1452 excreted in urine (Ae) | within 60 hours post-dose, depending on the assessment schedule for the cohort
  Categories: Placebo Tablet or Capsule, Placebo IV Solution, Debio 1450 IV solution, Debio 1450 Tablet, Debio 1450 Capsule, Debio 1450 oral solution
Percentage of cumulative amount of unchanged Debio 1450 and Debio 1452 excreted in urine (Ae%) | within 60 hours post-dose, depending on the assessment schedule for the cohort
  Categories: Placebo Tablet or Capsule, Placebo IV Solution, Debio 1450 IV solution, Debio 1450 Tablet, Debio 1450 Capsule, Debio 1450 oral solution
Renal clearance following oral administration | within 60 hours post-dose, depending on the assessment schedule for the cohort
  Categories: Placebo Tablet or Capsule, Debio 1450 Tablet, Debio 1450 Capsule, Debio 1450 oral solution

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Wittke, MD, Study Director — Debiopharm International SA
Locations (1):
- Early Phase Clinical Unit, Baltimore, Maryland, United States